CLINICAL TRIAL: NCT00095992
Title: A Phase II Study Of SB-715992 (NSC 727990) In Patients With Locally Advanced, Recurrent Or Metastatic Hepatocellular Carcinoma
Brief Title: SB-715992 in Treating Patients With Locally Advanced, Recurrent, or Metastatic Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I168; CAN-NCIC-IND168 (Other: PDQ); CDR0000391839 (Other: PDQ)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — ispinesib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: ispinesib — SB-715992 will be given as a 1 hour intravenous infusion in a dose of 18 mg/m2 once every 3 weeks

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as SB-715992, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well SB-715992 works in treating patients with locally advanced, recurrent, or metastatic liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of SB-715992, in terms of response rate and stable disease rate, in patients with locally advanced, recurrent, or metastatic hepatocellular carcinoma.
* Determine the toxicity of this drug in these patients.
* Determine the early progression rate and response duration in patients treated with this drug.
* Determine the pharmacokinetics of this drug in these patients.
* Correlate pharmacokinetics with safety and efficacy of this drug in these patients.
* Correlate tumor expression of β-tubulin and kinesin spindle protein with clinical outcomes in patients treated with this drug.

OUTLINE: This is a non-randomized, multicenter study.

Patients receive SB-715992 IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

All patients are followed at 4 weeks. Patients with ongoing stable or responding disease are followed every 3 months until relapse.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 12-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed hepatocellular carcinoma

  * Locally advanced, recurrent, or metastatic disease
  * Histologically confirmed disease must have archival paraffin-fixed tumor specimen available
* Measurable disease

  * At least 1 unidimensionally measurable site of disease ≥ 20 mm by x-ray, physical exam, or non-spiral CT scan OR ≥ 10 mm by spiral CT scan
  * Outside of previously irradiated area

    * Patients whose sole site of disease is in a previously irradiated field are eligible provided there is evidence of disease progression OR new lesions documented in the irradiated field
  * Bone metastases are not considered measurable disease
* Not curable by standard therapies
* No cholangiocarcinoma

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 80,000/mm^3

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST ≤ 5 times ULN
* Must have hepatic reserve of Child-Turcotte-Pugh class A or better

Renal

* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No myocardial infarction within the past 6 months
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No active cardiomyopathy
* No uncontrolled hypertension

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No clinical evidence of encephalopathy
* No ongoing or active infection
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to SB-715992
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No other malignancies within the past 5 years except adequately treated nonmelanoma skin cancer, curatively treated carcinoma in situ of the cervix, or other curatively treated solid tumors with no evidence of disease for at least 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since prior intra-hepatic chemotherapy as a component of trans-arterial chemoembolization and recovered

  * Documented disease progression
* No prior systemic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

  * Exceptions may be made for low-dose, nonmyelosuppressive radiotherapy

Surgery

* At least 4 weeks since prior major surgery
* Prior liver transplantation allowed

Other

* No other prior systemic therapy
* At least 4 weeks since prior local ablative therapy (e.g., radiofrequency ablation or ethanol injection) and recovered

  * Documented disease progression
* More than 28 days since prior investigational agents
* More than 14 days since prior and no concurrent use of any of the following CYP3A4 inhibitors or inducers:

  * Clarithromycin
  * Erythromycin
  * Troleandomycin
  * Itraconazole
  * Ketoconazole
  * Fluconazole (dose > 200 mg/day)
  * Voriconazole
  * Nefazodone
  * Fluvoxamine
  * Verapamil
  * Diltiazem
  * Grapefruit juice
  * Bitter orange
  * Phenytoin
  * Carbamazepine
  * Phenobarbital
  * Oxcarbazepine
  * Rifampin
  * Rifabutin
  * Rifapentine
  * Hypericum perforatum (St. John's wort)
  * Modafinil
* At least 6 months since prior and no concurrent amiodarone
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-03-08 (Actual); Primary Completion 2006-09-26 (Actual); Study Completion 2008-09-22 (Actual)

PRIMARY OUTCOMES:
Response | 4 years

SECONDARY OUTCOMES:
Toxicity | 4 years
Pharmacokinetics at day 1 of course 1 (day 1 of course 2 if dose is adjusted) | 4 years
Molecular correlates on archival tumor specimens and peripheral blood mononuclear cells (PBMCs) | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Knox, MD, Study Chair — Princess Margaret Hospital, Canada; Sharlene Gill, MD, Study Chair — British Columbia Cancer Agency
Locations (4):
- Canada (4):
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Knox JJ, Gill S, Synold TW, Biagi JJ, Major P, Feld R, Cripps C, Wainman N, Eisenhauer E, Seymour L. A phase II and pharmacokinetic study of SB-715992, in patients with metastatic hepatocellular carcinoma: a study of the National Cancer Institute of Canada Clinical Trials Group (NCIC CTG IND.168). Invest New Drugs. 2008 Jun;26(3):265-72. doi: 10.1007/s10637-007-9103-2. Epub 2008 Jan 15. PMID 18196204